CLINICAL TRIAL: NCT01718470
Title: Proseal Laryngeal Mask Airway Attenuates Systemic and Cerebral Hemodynamic Response During Awakening of Neurosurgical Patients
Brief Title: Proseal Laryngeal Mask Airway or Endotracheal Tube for Emergence From Neuroanesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ricard Valero (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, Ricard Valero, Ricard Valero M.D, Ph.D, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LMAvsETT
Record Dates: First submitted 2012-10-18; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension on Emergence
Keywords: Systolic blood pressure; Heart rate; Laryngeal mask; Endotracheal tube; craniotomy
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotracheal tube (Active Comparator): At the end of surgery, emerge from anesthesia with the ETT still in place
  Interventions: Procedure: Endotracheal tube
- Laryngeal mask (Active Comparator): At the end of surgery,emerge from anesthesia after ETT had been replaced by an LMA.
  Interventions: Procedure: LMA

INTERVENTIONS:
Procedure: Endotracheal tube — Hemodynamic variables were recorded at 8 moments: baseline, in the operating room one minute before anesthetic induction; 5 minutes after the end of surgery before awakening (ETT group) and 1, 5, 10, 15, 30 and 60 min after extubation . The last blood pressure and heart rate measurements were taken in the postoperative recovery room.
  Arms: Endotracheal tube
Procedure: LMA — Hemodynamic variables were recorded at 8 moments: baseline, in the operating room one minute before anesthetic induction; 5 minutes after the end of surgery before tube replacement (LMA group); and 1, 5, 10, 15, 30 and 60 min after LMA removal. The last blood pressure and heart rate measurements were taken in the postoperative recovery room.
  Other Names: Laryngeal mask
  Arms: Laryngeal mask

SUMMARY:
Extubation and emergence from anesthesia lead to systemic and cerebral hemodynamic changes that can cause cerebral edema and hemorrhage. The hemodynamic profile on emergence is more favorable if a laryngeal mask airway (LMA) is inserted before neurosurgical patients emerge from anesthesia. We aimed to compare the impact of awakening neurosurgery patients after insertion of a ProSeal LMA to replace the endotracheal tube (ETT).

DETAILED DESCRIPTION:
At the end of surgery, the anesthesiologist opened a sealed envelope labeled with software-generated randomized numbers to learn the patient's assignment to one of two groups to emerge from anesthesia with the ETT still in place or after it had been replaced by an LMA.

Hemodynamic variables were recorded at 8 moments: baseline, in the operating room one minute before anesthetic induction; 5 minutes after the end of surgery before awakening (ETT group) or before tube replacement (LMA group); and 1, 5, 10, 15, 30 and 60 min after extubation or LMA removal (according to group assignment).

ELIGIBILITY:
Inclusion Criteria:

* Elective craniotomy

Exclusion Criteria:

* Difficult airway
* Uncontrolled hypertension before surgery
* gastroesophageal reflux

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure change | 1 minute before anesthesia induction, 5 minutes before extubation, and minute 1, 5, 10, 15, 30 and 60 after extubation

SECONDARY OUTCOMES:
heart rate change | 1 minute before anesthesia induction, 5 minutes before extubation, and minutes 1,5,10,15,30 and 60 after extubation

OTHER OUTCOMES:
Norepinephrine plasma concentration change | 1 minute before anesthesia induction, 1 minute and 30 minutes after extubation,

CONTACTS AND LOCATIONS:
Overall Officials: Perelló Laura, MD, Principal Investigator — Anesthesia Specialist, Anesthesia department, Hospital Clínic de Barcelona
Locations (1):
- Anesthesia department, Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Bruder N, Stordeur JM, Ravussin P, Valli M, Dufour H, Bruguerolle B, Francois G. Metabolic and hemodynamic changes during recovery and tracheal extubation in neurosurgical patients: immediate versus delayed recovery. Anesth Analg. 1999 Sep;89(3):674-8. doi: 10.1097/00000539-199909000-00027. PMID 10475304